CLINICAL TRIAL: NCT07014007
Title: Open-label Study to Assess the Tolerance and Efficacy of the Product RV4421B-EV0407, Applied in Paediatric and Adult Populations With Mild to Moderate Atopic Dermatitis for 12 Weeks
Brief Title: Tolerance and Efficacy Open-label Study With RV4421B, in Various Populations With Atopic Dermatitis for 12 Weeks
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV44221B20240736
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema; Flare; Inflammatory skin disease; Altered skin barrier; Dryness; Itching; Redness; Stinging; Burning sensation
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Pruritus; Erythema; Paresthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infant group (Experimental): Subjects aged from 3 months to 23 months old included
  Medical device: RV4421B- EV0407 the test product will be applied twice daily alone or in association with topical corticosteroids.
  Interventions: Device: RV4421B- EV0407
- Children group (Experimental): Subjects aged from 24 months to 12 years old included
  Medical device: RV4421B- EV0407 the test product will be applied twice daily alone or in association with topical corticosteroids.
  Interventions: Device: RV4421B- EV0407
- Teenagers & adults group (Experimental): Subjects aged from 13 years old
  Medical device: RV4421B- EV0407 the test product will be applied twice daily alone or in association with topical corticosteroids.
  Interventions: Device: RV4421B- EV0407

INTERVENTIONS:
Device: RV4421B- EV0407 — Medical device. Product application on studied areas, 5 to 15 minutes after corticosteroids application, if applicable. The maximum duration of application of medical device is 87 days.

SUMMARY:
Pierre Fabre Laboratories have developed a cream with medical device status, RV4421B-EV0407 indicated for the treatment of eczemas, including atopic eczema, contact eczema and chronic hand eczema.

This product is already marketed in several countries. The objective of this clinical study is to evaluate the safety and efficacy of the study product when used alone or in association with topical corticosteroid therapy, in an ethnically diverse adult and pediatric population (including dark skin) and over a long period of time with a 12-week follow-up.

5 visits are planned:

* Visit 1: Inclusion visit (Day 1)
* Visit 2: Intermediate visit (Phone visit - Between Day 8 and Day 15)
* Visit 3: Intermediate visit (Day 29 ± 3 days)
* Visit 4: Intermediate visit (Day 57 ± 3 days)
* Visit 5: End of study visit (Day 85 ± 3 days)

ELIGIBILITY:
Inclusion criteria:

* Male or female, with any phototype according to Fitzpatrick classification aged:
* Group 1 (infants group): from 3 months to 23 months old included
* Group 2 (children group): from 24 months to 12 years old included
* Group 3 (teenagers & adults group): from 13 years old
* Subject with a diagnosis of atopic dermatitis according to the U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis (Williams HC, Burney PG, et al.).
* Subject with studied areas (lesions and prevailing xerotic areas) limited up to 30% of the body surface area
* Subject with mild to moderate Atopic Dermatitis

Criteria related to treatments and/or products:

• Topical corticosteroids treatments (following international treatment guidelines for each age sub-group and including investigator agreement) applied on AD lesions areas since 1 to 5 days before the inclusion and ongoing at the time of inclusion. *

*The investigator will be authorized to adjust the treatment during the study.

Exclusion criteria:

Criteria related to the skin condition or the disease:

* Infant with Atopic Dermatitis lesions or prevailing xerotic areas located on the diaper (groups 1 & 2)
* Subject with history of allergy or intolerance to any of the study product(s) ingredients or material used for the research
* Subject having any other dermatologic condition than Atopic Dermatitis, or characteristics (like tattoo…) on the studied areas liable to interfere with the study assessments
* Subject having a dermatological condition, an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Knowledge of Acquired Immunodeficiency Syndrome or Infectious (acute or chronic)

Criteria related to treatments and/or products:

* Systemic biological immunosuppressive treatment established or modified within 12 weeks before the inclusion or planned to be started during the study
* Phototherapy performed within 4 weeks before the inclusion visit or planned to be started during the study
* Systemic non-biological immunosuppressive treatment established or modified within 4 weeks before the inclusion or ongoing or planned to be started during the study
* Systemic corticosteroids treatment established or modified within 4 weeks before the inclusion or ongoing or planned to be started during the study
* Systemic antibiotics for dermatological purposes treatment established or modified within 2 weeks before the inclusion or ongoing or planned to be started during the study
* Systemic antihistaminic treatment established or modified within 2 weeks before the inclusion
* Topical treatments (immunomodulators (TIMs), non-steroidal anti-inflammatory, antihistaminic, antibiotics for dermatological purposes or antiseptics) applied on studied areas within 1 week before the inclusion or ongoing or planned to be started during the study
* Any other topical treatment or product applied on studied areas incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Skin care product (including moisturizer) applied on the whole body between the evening before the visit and the inclusion.
* Water and/or any cleansing product, applied on the whole body within 4 hours before the inclusion visit. If there is no studied area on the face, the subject is allowed to do a light face wash without time restriction (especially in the morning of the visit).
* Subject who plans to modify his/her usual moisturizer (allowed outside studied areas) and/or care habits during the study

Treatment of the mother if the subject of group 1 and 2 is breastfed:

* Systemic biological immunosuppressive treatment established or modified within 12 weeks before the inclusion or planned to be started during the study
* Systemic non-biological immunosuppressive treatment established or modified within 4 weeks before the inclusion or planned to be started during the study
* Systemic corticosteroids established or modified within 2 weeks before the inclusion or planned to be started during the study
* Systemic antihistaminic established or modified within 2 weeks before the inclusion
* Systemic antibiotics for dermatological purposes established or modified within 1 week before the inclusion or planned to be started during the study

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Local tolerance of the product RV4421B-EV0407 on studied areas | Day 85
  The results of the local tolerance will take into account the clinical signs observed by the investigators and the signs reported by the subject and/or the subjects' parent(s) or guardian(s), based on a 5-point scale (From 1 = Excellent tolerance to 5 = Bad tolerance)

SECONDARY OUTCOMES:
Local tolerance of the product RV4421B-EV0407 on studied areas at several timepoints | Day 1, 10 to 30 minutes after the first application, Day 29 & Day 57
  using the same 5-point scale as the primary criterion and same rules.
Recording of adverse events | From Day 1 to Day 85
  At each visit, the occurrence of Adverse Events since the last visit will be determined by the subject's / parent(s) or guardian(s) spontaneous reporting, the investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the CRF
Local-SCORAD (SCORing Atopic Dermatitis) | Day 1, Day 29, Day 57 & Day 85
  Local -SCORAD (SCORing Atopic Dermatitis) will be assessed by the investigator on target area (= area most representative of Atopic Dermatitis severity of the whole body) on a scale ranged from 0 to 15, at each visit (except the Visit 2).
  Each of 5 objective signs of the SCORAD (Erythema, Oedema/papulation, Oozing/Crusts, Excoriation, and Lichenification) will be rated from 0 (absent) to 3 (severe) independently
SCORAD (SCORing Atopic Dermatitis) | Day 1, Day 29, Day 57 & Day 85
  SCORAD will be assessed by the investigator at each visit (except the Visit 2). The SCORAD is a scoring system based on the assessment of extent and intensity in a standardized manner. The complete system is called SCORAD index and takes into account the extent of the lesions, the severity of the clinical signs (objective signs) and the subjective symptoms (pruritus, sleep loss) reported on a Visual Analogue Scale (VAS).
  The extent of lesions is scored on an evaluation form. The intensity is determined by grading each of the six items on a scale from 0 to 3 (erythema, oedema/papulation, oozing/crusts, excoriation, lichenification and dryness). Each item should be scored on the most representative area for a given intensity item.
IGA (Investigator's Global Assessment) | Day 1, Day 29, Day 57 & Day 85
  IGA (Investigator's Global Assessment) will be assessed by the investigator on a 6-point scale ranged from 0 (= clear) to 5 (=very severe disease), at each visit (except the Visit 2).
PO-SCORAD (Patient Oriented SCORing Atopic Dermatitis) | Every 2 weeks ± 2 days (or during the visit at site for sequences close to visit at site) from Day 1 to Day 85
  PO-SCORAD (Patient Oriented SCORing Atopic Dermatitis) will be assessed by the subject / subject's parent(s) or guardian(s) every 2 weeks* from Day 1 to Day 85 (± 3 days) The PO-SCORAD index and each of its intensity items components will be assessed on a scale ranged from 0 to 3 (0=none; 1=mild; 2=moderate; 3=severe).
  The PO-SCORAD is composed of 3 parts:
  * Part 1: Extent: Surface area of skin affected by eczema (drawing/colouring the infected area on a scheme)
  * Part 2 : Objective signs:
    * Evaluation on a 4-point scale (from 0 (=none) to 3(=severe) of the dryness of the skin without eczema
    * Evaluation on a 4-point scale (from 0 (=none) to 3(=severe) of the severity of the eczema: redness of the skin affected by eczema, swelling, oozing/crust, scratching and thickening
  * Part 3 : Subjective symptoms (evaluation of the sleep disturbance and the itching)
SGA (Subject's Global Assessment) | Every 2 weeks ± 2 days (or during the visit at site for sequences close to visit at site) from Day 15 to Day 85
  SGA (Subject's Global Assessment) will be assessed by the subject / subject's parent(s) or guardian(s) on a 5-point scale ranged from -2 (=Significant worsening) to +2 (=Significant improvement), every 2 weeks in comparison to Atopic Dermatitis intensity baseline: Day 1.
Subject quality of life DLQI for subjects from 16 years | Every 4 weeks ± 2 days (or during the visit at site for sequences close to visit at site) from Day 29 to Day 85
  Subject quality of life will be assessed by the subject by means of the Dermatology Life Quality Index (DLQI) questionnaire every 4 weeks
  This questionnaire of quality of life is designed to be completed with a one-week recall period. It is calculated by summing the score of 10 questions, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Subject quality of life CDLQI for subjects from 4 years to 15 years included | Every 4 weeks ± 2 days (or during the visit at site for sequences close to visit at site) from Day 29 to Day 85
  Subject quality of life will be assessed by the subject by means of the Children's Dermatology Life Quality Index (CDLQI) questionnaire every 4 weeks
  This questionnaire of quality of life is designed to be completed with a one-week recall period. It is calculated by summing the score of 10 questions, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Subject quality of life IDQOL for subjects from 3 months to 3 years included | Every 4 weeks ± 2 days (or during the visit at site for sequences close to visit at site) from Day 29 to Day 85
  Subject quality of life will be assessed by the subject by means of the Infant Dermatology Quality of Life Index (IDQOL) questionnaire every 4 weeks
  This questionnaire of quality of life is designed to be completed with a one-week recall period. It is calculated by summing the score of 10 questions, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Subject's satisfaction questionnaire | at Day 1 (10 to 30 minutes after the 1st product application), within 2 days before Day 29 or at Day 29 (± 3 days), within 2 days before Day 85 or at Day 85 (± 3 days)
  Satisfaction as regards to the use of the test product will be assessed by the subject / subject's parent(s) or guardian(s) through a specific questionnaire.